CLINICAL TRIAL: NCT00198380
Title: Phase II of Gefitinib (IRESSA) Administered as First-line Treatment in Patients With Non-resectable Pneumonic-type Adenocarcinoma (P-ADC)
Brief Title: Treatment of Lung Adenocarcinoma With Bronchioloalveolar Feature
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0401
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Pneumonic-type Adenocarcinoma (P-ADC); Lung Adenocarcinoma With Bronchiolo-alveolar Feature
Keywords: Adenocarcinoma, Bronchiolo-Alveolar
MeSH Terms: conditions — Adenocarcinoma, Bronchiolo-Alveolar | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250 mg/day, until progression or severe toxicity

SUMMARY:
Pneumonic adenocarcinoma (P-ADC) is defined as a primary lung ADC with a radiological pneumonic presentation, usually referred to histologically as ADC with a mixed-invasive and BAC predominant subtype in the 2004 WHO classification. Surgery is the best therapy for resectable tumors since the effectiveness of chemotherapy is disappointing. In the advanced P-ADC diffuse/multifocal types of BAC, epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) (gefitinib and erlotinib) have shown promise, with some rapid, dramatic responses, possibly reflecting specific molecular differences from other non-small cell lung carcinomas.

DETAILED DESCRIPTION:
We therefore conducted a French multicentric phase II trial (IFCT 0401) to evaluate activity and tolerance of gefitinib (250 mg/day) administered as first line treatment in patients with non-resectable P-ADC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically / cytologically proven ADC-P
* Non-resectable disease
* 3-month expected survival
* No prior radiotherapy or chemotherapy
* Age >= 18 years old
* Performance status < 4 (WHO)
* Adequate blood biological parameters

Exclusion Criteria:

* Abnormal initial fibroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Disease control rate after 3 months of treatment | Month

SECONDARY OUTCOMES:
Quality of life | 3-month
Time to progression | month
Survival | month
Prediction disease control by clinical and biological markers | month

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Cadranel, Pr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (11):
- France (11):
  - CHU Besancon - Pneumologie, Besançon
  - APHP - CHU Avicenne - Oncologie Medicale, Bobigny
  - Centre F. Baclesse, Caen
  - CHU - Pneumologie, Caen
  - CHU Grenoble - pneumologie, Grenoble
  - HCL - Croix-Rousse, Lyon
  - APHP - Saint-Antoine - pneumologie, Paris
  - Hopital Tenon - Pneumologie, Paris
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - CHU Saint-Etienne Pneumologie, Saint-Etienne
  - CHU Lyautey - Pneumologie, Strasbourg

REFERENCES:
- [Background] Cadranel J, Lavole A, Gounant V, Wislez M. [Bronchioloalveolar carcinoma and adenocarcinoma with bronchioloalveolar features: a clinico-pathological spectrum]. Rev Mal Respir. 2007 Oct;24(8 Pt 2):6S165-70. French. PMID 18235410
- [Background] Wislez M, Massiani MA, Milleron B, Souidi A, Carette MF, Antoine M, Cadranel J. Clinical characteristics of pneumonic-type adenocarcinoma of the lung. Chest. 2003 Jun;123(6):1868-77. doi: 10.1378/chest.123.6.1868. PMID 12796162
- [Background] Garfield DH, Cadranel JL, Wislez M, Franklin WA, Hirsch FR. The bronchioloalveolar carcinoma and peripheral adenocarcinoma spectrum of diseases. J Thorac Oncol. 2006 May;1(4):344-59. PMID 17409882
- [Result] Cadranel J, Quoix E, Baudrin L, Mourlanette P, Moro-Sibilot D, Morere JF, Souquet PJ, Soria JC, Morin F, Milleron B; IFCT-0401 Trial Group. IFCT-0401 Trial: a phase II study of gefitinib administered as first-line treatment in advanced adenocarcinoma with bronchioloalveolar carcinoma subtype. J Thorac Oncol. 2009 Sep;4(9):1126-35. doi: 10.1097/JTO.0b013e3181abeb5d. PMID 19574932
- [Result] Wislez M, Antoine M, Baudrin L, Poulot V, Neuville A, Pradere M, Longchampt E, Isaac-Sibille S, Lebitasy MP, Cadranel J. Non-mucinous and mucinous subtypes of adenocarcinoma with bronchioloalveolar carcinoma features differ by biomarker expression and in the response to gefitinib. Lung Cancer. 2010 May;68(2):185-91. doi: 10.1016/j.lungcan.2009.05.021. Epub 2009 Jul 5. PMID 19581016
- See also: Official website — http://www.ifct.fr